CLINICAL TRIAL: NCT03669952
Title: Longitudinal Observational Study About the Influence of Ductal Carcinoma in Situ on the Outcome of Invasive Breast Cancer
Brief Title: Study of the Influence of Ductal Carcinoma in Situ on the Outcome of Invasive Breast Cancer
Status: Completed | Type: Observational
Sponsor: Omphis Foundation (Other)
Responsible Party: Principal Investigator, Sandra Lopez Gordo, Specialists in General Surgery, Omphis Foundation
Other Study IDs: SLG_01
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Outcome of Breast Cancer
Keywords: Breast cancer; Ductal carcinoma in situ; Invasive ductal carcinoma; Prognosis factors
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Invasive ductal carcinoma: Patients with Invasive ductal carcinoma
  Interventions: Other: None intervention

INTERVENTIONS:
Other: None intervention — No interventions are realized, only observational study

SUMMARY:
A prospective observational longitudinal study of 464 patients was performed between 2010 and 2015. Patients with invasive ductal carcinoma (IDC) and ductal carcinoma in situ associated to invasive ductal carcinoma (DCIS +IDC) were included and analyzed.

DETAILED DESCRIPTION:
Type of study:

A prospective observational longitudinal study was performed on patients who had undergone curative surgery for primary invasive breast cancer between 2010 and 2015. The study was performed in a single breast pathology unit [Alt Penedés hospital and Sant Camil hospital(GAP)]. Only patients with a definitive histopathology-based diagnostic of ductal carcinoma were included. Patients diagnosed with metastasis were excluded. Patients with bilateral breast cancer were included as two independent study cases.

Patients:

Sample size calculation: 191. A total of 464 patients were included in the study. IDC was present in 221 patients (47.6%) and IDC + DCIS was present in 243 patients (52.4%).

Data collected included clinical characteristics (age, laterality and clinical symptoms at the time of diagnostic), histopathological information (tumor size, tumor grade, hormone receptors, nodal status, HER-2 mutation (erb-b2 receptor tyrosine kinase 2), number of ki67, presence and percentage of DCIS, grade of DCIS, and surrogate subtype) and surgical procedure performed.

Tumor histopathology and the number of lymph nodes involved were evaluated by routine hematoxylin-eosin (H&E) staining. The histological response to chemotherapy was assessed according to Miller-Payne criteria of grading (MPG) and Residual Disease in Breast and Nodes (RDBN).

The percentage of DCIS and its grade (classified as low, intermediate or high) was measured by two independent pathologists.

Statistical analysis:

Quantitative data are shown as the median or mean of values and their variability is expressed as the range or standard deviation (SD), as specified for each analysis. Qualitative data are shown as absolute values or percentages. The incidence was used as a measure of frequency and the relative risk as a measure of association between independent groups.

The study of the normality of quantitative variables was done applying the Kolmogorov-Smirnov or the Shapiro-Wilk tests, as indicated for each analysis. For significance assessment of quantitative data, unpaired Student's T-test or two-tailed Mann-Whitney U test was applied, as specified for each analysis. For significance assessment of qualitative data, Fisher's exact test or Chi-squared test was applied. For the analysis of more than two groups, one-way ANOVA and Tukey's range test for post hoc pairwise comparison of groups, or Kruskal-Wallis were used. Survival was analyzed with the Kaplan-Meier estimate and survival distributions compared with the Log-Rank test. Multivariate Cox proportional hazards regression model was used to simultaneously evaluate the effect of several factors on survival and mortality.

Statistical analysis was performed using the software SPSS® (Statistical Package for the Social Sciences) version 21.

The aim of the investigator's study is to compare the clinical and histopathological factors between patients with IDC or DCIS-associated IDC (IDC + DCIS) and find the prognostic factors associated to recurrence and mortality in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with invasive ductal carcinoma of the breast
* Patients who received surgery for primary invasive breast cancer between 2010 and 2015

Exclusion Criteria:

* Patients with metastasis at the diagnostic

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population included in the study was 464 patients. IDC was present in 221 patients (47.6%) and IDC + DCIS was present in 243 patients (52.4%).
Sampling Method: Probability Sample
Enrollment: 464 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Recurrence | Patients included between 2010 and 2015 will be follow up til January of 2018 with a mean follow up of 51.43 months
  Neoplasm metastasis, either local or distant recurrence of the invasive ductal carcinoma

IPD SHARING:
Plan to Share IPD: No